Prospective, Randomized, Fellow Eye-Controlled Study of Postoperative Pain and Inflammation Control with an Intracanalicular Dexamethasone 0.4 mg Ophthalmic Insert Following Small Incision Lenticule Extraction

22NOVEMBER2022

NCT04380857

## Statistical Analysis Plan: No formal power analysis was conducted, and the sample size was set at 40 eyes based on the sample size used in several similar prior studies.18–20 Chi-square tests were used to compare proportions and t-tests to compare means. The level of significance was set at 0.05.